CLINICAL TRIAL: NCT02387515
Title: Technology-supported Exercise Therapy for Patients With Chronic Low Back Pain: Pilot Study
Brief Title: Technology-supported Exercise Therapy for Patients With Chronic Low Back Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hasselt University (Other)
Collaborators: Jessa Hospital (Other)
Responsible Party: Principal Investigator, Annick Timmermans, prof. dr., Hasselt University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: PILOT2013TM01
Record Dates: First submitted 2014-12-13; First posted 2015-03-13 (Estimated); Last update posted 2017-08-09 (Actual); Status verified 2017-08

CONDITIONS: Chronic Non-specific Low Back Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- intensive rehabilitation program (Experimental): Patients will follow an intensive rehabilitation program (2x/week for 18 weeks), with emphasis on motor control training that is supported by technology.
  Interventions: Other: intensive rehabilitation program

INTERVENTIONS:
Other: intensive rehabilitation program — Patients will follow an intensive rehabilitation program (2x/week for 18 weeks), with emphasis on motor control training that is supported by technology. The technological system consists out of motion tracking sensors that register the movements and position of the lumbar spine.

SUMMARY:
This clinical pilot trial will investigate the effects of technology-supported exercise therapy for chronic non-specific low back pain. Patients will follow an intensive rehabilitation program (2x/week for 18 weeks), with emphasis on motor control training that is supported by technology. The technological system consists out of motion tracking sensors that register the movements and position of the lumbar spine.

ELIGIBILITY:
Inclusion Criteria:

* 18-65 y.o.
* Chronic non-specific low back pain, with or without leg pain
* Motor control impairment
* Sufficient knowledge of the Dutch language to understand instructions

Exclusion Criteria:

* Spinal surgery in the past
* Underlying serious pathologies (tumor, fracture, neurological diseases)
* Signs or symptoms of nerve root compression
* Pregnancy or less than 1 year post-partum
* Known allergy for tape

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2013-12; Primary Completion 2015-03 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
The numeric pain rating scale | baseline
  the numeric pain rating scale (0-10)
The numeric pain rating scale | week 3
  the numeric pain rating scale (0-10)
The numeric pain rating scale | week 8
  the numeric pain rating scale (0-10)months post-intervention.
The numeric pain rating scale | week 13
  the numeric pain rating scale (0-10)
The numeric pain rating scale | week 18
  the numeric pain rating scale (0-10)
The numeric pain rating scale | week 44
  the numeric pain rating scale (0-10)
Roland Morris Questionnaire (0-24) | baseline
  Roland Morris Questionnaire (0-24)
Roland Morris Questionnaire (0-24) | week 3
  Roland Morris Questionnaire (0-24)
Roland Morris Questionnaire (0-24) | week 8
  Roland Morris Questionnaire (0-24)
Roland Morris Questionnaire (0-24) | week 13
  Roland Morris Questionnaire (0-24)
Roland Morris Questionnaire (0-24) | week 18
  Roland Morris Questionnaire (0-24)
Roland Morris Questionnaire (0-24) | week 44
  Roland Morris Questionnaire (0-24)
Patient specific functioning scale (0-10) | baseline
  Patient specific functioning scale (0-10)
Patient specific functioning scale (0-10) | week 3
  Patient specific functioning scale (0-10)
Patient specific functioning scale (0-10) | week 8
  Patient specific functioning scale (0-10)
Patient specific functioning scale (0-10) | week 13
  Patient specific functioning scale (0-10)
Patient specific functioning scale (0-10) | week 18
  Patient specific functioning scale (0-10)
Patient specific functioning scale (0-10) | week 44
  Patient specific functioning scale (0-10)
Pain self-efficacy questionnaire (0-60) | baseline
  Pain self-efficacy questionnaire (0-60)
Pain self-efficacy questionnaire (0-60) | week 3
  Pain self-efficacy questionnaire (0-60)
Pain self-efficacy questionnaire (0-60) | week 8
  Pain self-efficacy questionnaire (0-60)
Pain self-efficacy questionnaire (0-60) | week 13
  Pain self-efficacy questionnaire (0-60)
Pain self-efficacy questionnaire (0-60) | week 18
  Pain self-efficacy questionnaire (0-60)
Pain self-efficacy questionnaire (0-60) | week 44
  Pain self-efficacy questionnaire (0-60)
the Tampa scale for kinesiophobia (17-68) | baseline
  the Tampa scale for kinesiophobia (17-68)
the Tampa scale for kinesiophobia (17-68) | week 3
  the Tampa scale for kinesiophobia (17-68)
the Tampa scale for kinesiophobia (17-68) | week 8
  the Tampa scale for kinesiophobia (17-68)
the Tampa scale for kinesiophobia (17-68) | week 13
  the Tampa scale for kinesiophobia (17-68)
the Tampa scale for kinesiophobia (17-68) | week 18
  the Tampa scale for kinesiophobia (17-68)
the Tampa scale for kinesiophobia (17-68) | week 44
  the Tampa scale for kinesiophobia (17-68)
Patient satisfaction with treatment (0-10) | baseline
  Patient satisfaction with treatment (0-10)
Patient satisfaction with treatment (0-10) | week 3
  Patient satisfaction with treatment (0-10)
Patient satisfaction with treatment (0-10) | week 8
  Patient satisfaction with treatment (0-10)
Patient satisfaction with treatment (0-10) | week 13
  Patient satisfaction with treatment (0-10)
Patient satisfaction with treatment (0-10) | week 18
  Patient satisfaction with treatment (0-10)
Patient satisfaction with treatment (0-10) | week 44
  Patient satisfaction with treatment (0-10)

SECONDARY OUTCOMES:
short form 36 | baseline
  Quality of life, SF-36 questionnaire
short form 36 | week 3
  Quality of life, SF-36 questionnaire
short form 36 | week 8
  Quality of life, SF-36 questionnaire
short form 36 | week 13
  Quality of life, SF-36 questionnaire
short form 36 | week 18
  Quality of life, SF-36 questionnaire
short form 36 | week 44
  Quality of life, SF-36 questionnaire
Credibility and expectancy questionnaire | baseline
  Credibility and expectancy questionnaire
Credibility and expectancy questionnaire | week 3
  Credibility and expectancy questionnaire
Credibility and expectancy questionnaire | week 8
  Credibility and expectancy questionnaire
Credibility and expectancy questionnaire | week 13
  Credibility and expectancy questionnaire
Credibility and expectancy questionnaire | week 18
  Credibility and expectancy questionnaire
Credibility and expectancy questionnaire | week 44
  Credibility and expectancy questionnaire
Intrinsic motivation inventory form | baseline
  Intrinsic motivation inventory form
Intrinsic motivation inventory form | week 3
  Intrinsic motivation inventory form
Intrinsic motivation inventory form | week 8
  Intrinsic motivation inventory form
Intrinsic motivation inventory form | week 13
  Intrinsic motivation inventory form
Intrinsic motivation inventory form | week 18
  Intrinsic motivation inventory form
Work absenteeism because of LBP (low back pain) (yes (% of absenteeism), no) | baseline
  Work absenteeism because of LBP (low back pain) (yes (% of absenteeism), no)
Work absenteeism because of LBP (low back pain) (yes (% of absenteeism), no) | week 3
  Work absenteeism because of LBP (low back pain) (yes (% of absenteeism), no)
Work absenteeism because of LBP (low back pain) (yes (% of absenteeism), no) | week 8
  Work absenteeism because of LBP (low back pain) (yes (% of absenteeism), no)
Work absenteeism because of LBP (low back pain) (yes (% of absenteeism), no) | week 13
  Work absenteeism because of LBP (low back pain) (yes (% of absenteeism), no)
Work absenteeism because of LBP (low back pain) (yes (% of absenteeism), no) | week 18
  Work absenteeism because of LBP (low back pain) (yes (% of absenteeism), no)
Work absenteeism because of LBP (low back pain) (yes (% of absenteeism), no) | week 44
  Work absenteeism because of LBP (low back pain) (yes (% of absenteeism), no)
Adherence to exercise program assessed by number of visits attended and self-reported adherence to home exercises | baseline
  Adherence to exercise program (number of visits attended, self-reported adherence to home exercises)
Adherence to exercise program assessed by number of visits attended and self-reported adherence to home exercises | week 3
  Adherence to exercise program (number of visits attended, self-reported adherence to home exercises)
Adherence to exercise program assessed by number of visits attended and self-reported adherence to home exercises | week 8
  Adherence to exercise program (number of visits attended, self-reported adherence to home exercises)
Adherence to exercise program assessed by number of visits attended and self-reported adherence to home exercises | week 13
  Adherence to exercise program (number of visits attended, self-reported adherence to home exercises)
Adherence to exercise program assessed by number of visits attended and self-reported adherence to home exercises | week18
  Adherence to exercise program (number of visits attended, self-reported adherence to home exercises)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Matheve, drs., Study Chair — Hasselt University; annick Timmermans, prof.dr., Principal Investigator — Hasselt University; Guido Claes, MD, Study Chair — Jessa Hospital
Locations (1):
- Universiteit Hasselt, Hasselt, Belgium